CLINICAL TRIAL: NCT03439176
Title: A Pilot Evaluation Exploring New Adhesive Materials and Their Ability to Handle Moisture From Abdominal and Peristomal Skin
Brief Title: Investigating the Adhesion of New Adhesive to the Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP267_3_5
Record Dates: First submitted 2018-01-31; First posted 2018-02-20 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of new adhesive strips (Experimental): The subjects will test adhesives strips made of 4 different adhesives:
  Standard adhesive 1 Standard adhesive 2 PL4 PL16-L
  Interventions: Other: Standard adhesive 1; Other: Standard adhesive 2; Other: PL4; Other: PL16-L

INTERVENTIONS:
Other: Standard adhesive 1 — This strip contains a standard hydrocolloid adhesive found in ostomy devices
Other: Standard adhesive 2 — This strip contains a standard hydrocolloid adhesive found in ostomy devices
Other: PL4 — This strip contains a new adhesive
Other: PL16-L — This strip contains a new adhesive

SUMMARY:
The adhesion of the new adhesive strips is investigated on healthy volunteers

DETAILED DESCRIPTION:
Inclusion visit:

* Introduction to the study
* Inclusion in study
* Baseline information is obtained
* Instruct subject to pre-strip of abdominal skin

Test visits 1-25 (up to maximum 25 visits per subject. (1-3 days after pre-stripping the abdominal skin):

* Baseline measurements are conducted on both sides of the stomach (TEWL, hydration, erythema, pH - 3 repeated measurements under each adhesive strip area (upper, middle and bottom of adhesive strip)
* Potential wetting of skin - shower/bicycle exercise (max 60 minutes) and after-wetting baseline measurements are conducted (TEWL, hydration, erythema, pH - 3 times/strips (upper, middle and bottom of adhesive strip))
* Adhesive strips are weighted and applied
* Potential shower/bicycle exercise (max 60 minutes)
* Adhesive strips are removed at pre-defined timeslots (peel force measured)
* Discomfort when strip was peeled of is evaluated by subject (VAS)
* Measurements are conducted (TEWL, hydration, erythema, pH - 3 times/strips (upper, middle and bottom of adhesive strip))
* Acclimatization ½
* Measurements are conducted (TEWL, hydration, erythema, pH - 3 times/strips (upper, middle and bottom of adhesive strip))
* Adhesive strips are weighed
* Photo of adhesive strips

The subjects can be asked to apply and change strips every 24 hours between two test visits but for a maximum of 10 days between two visits. The strips should be applied at the same place every time.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have intact skin on the area used in the investigation

Exclusion Criteria:

1. Currently receiving or have within the past 2 months received radio- and/or chemotherapy
2. Currently receiving or have within the past months received topical steroid treatment in the abdominal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Have dermatological problems in the abdominal area (assessed by investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Swelling of the adhesive | 24 hours
  Swelling of adhesive strips measured by weight (difference between the weight of the strip before and after use)

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, Principal Investigator — Head of the pre-clinical department
Locations (1):
- Coloplast A/S, Humlebæk, Denmark